CLINICAL TRIAL: NCT02102997
Title: Deutsches Dual Therapy Stent Register
Acronym: DTS Register
Status: Terminated | Type: Observational
Why Stopped: Low enrolment
Sponsor: OrbusNeich (Industry)
Responsible Party: Sponsor
Other Study IDs: DTS.DE Register V 1.2
Record Dates: First submitted 2014-03-24; First posted 2014-04-03 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease
Keywords: DTS; Stents; Stent; DES; Drug eluting; Drug Eluting Stent (DES); Drug eluting stents; Endothelial Progenitor Cell (EPC); Endothelial progenitor cell capturing; Sirolimus; Sirolimus eluting; Percutaneous Coronary Intervention (PCI); PCI; Registry; Registries; Multi center; Multi centre
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The DTS.DE registry is an initiative for the collection of high quality process and historical data of implantations with the COMBO Dual Therapy Stent in Germany. DTS.DE was designed as a national, non- randomized, prospective, multicenter registry without a comparison group.

The responsible Steering Committee is of the opinion that the Combo stent qualifies for further documentation of treatment results in the form of a German registry, based the CE certification of the COMBO Dual Therapy stent in 2013 and its clinical and scientific investigation in the context of the REMEDEE study program, as well as company independent externally initiated studies with the COMBO Dual Therapy Stent.

It is expected that by mid- 2015, at least 1,000 patients will be enrolled and documented in the DTS.DE registry with the COMBO Dual Therapy Stent. A clinical follow-up is performed after 6 weeks and 12 months.

DETAILED DESCRIPTION:
It is the objective of the DTS.DE registry to capture the documentation of all patients who have been treated with a Combo Dual Therapy Stent in Germany, and who have been properly informed and consented with regards to their participation in the registry. All of these patients will be registered in the electronic data capturing system (eCRF) of the DTS.DE registry and will be followed and documented for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients has at least one coronary lesion, suitable for PCI treatment with the Combo stent in accordance with European Society of Cardiology Guidelines and local Guidelines of the Deutsche Gesellschaft für Kardiologie for drug eluting stents

Exclusion Criteria:

* Patient has previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti- Murine Antibodies (HAMA)
* Patient in whom anti-platelet and/or anticoagulant therapy is contraindicated
* Patient in whom a complete inflation of the angioplasty balloon or correct stent placement is thought to be inhibited

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Germany who have undergone PCI with the COMBO Dual Therapy Stent.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2013-07; Primary Completion 2017-08-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months
  TVF is defined as the hierarchical composite of target vessel related Major Adverse Cardiac Events (MACE). MACE is defined as the composite of death, myocardial infarction and target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Procedural success | Day of procedure
  Successful implantation of the stent and a residual stenosis of less than 20%
MACE | 6 weeks and 12 months
  MACE is defined as the composite of of death, myocardial infarction and target lesion revascularization
Stent induced serious adverse events (SAE) | 12 months
Stent thrombosis | 12 months
  Classified per ARC definitions as definite, probable or possible stent thrombosis
Thrombolysis in Myocardial Infarction (TIMI) bleeding | 12 months
  Bleeding as defined by the TIMI criteria: major, minor or minimal

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD, PhD, Study Director — Universitätsklinikum Ulm, Klinik für Innere Medizin II Albert-Einstein-Allee 23, 89081 Ulm, Germany; Michael Haude, MD, PhD, Study Director — Kardiologie Lukaskrankenhaus Neuss Preußenstraße 84 D-41464 Neuss, Germany; Bernward Lauer, MD, PhD, Study Director — Klinik für Kardiologie, Zentralklinik Bad Berka GmbH, Robert-Koch-Allee 9 99437 Bad Berka, Germany; Volker Schächinger, MD, PhD, Study Director — Kardiologie, Angiologie, Pneumologie, Intensivmedizin Klinikum Fulda gAG Pacelliallee 4 - 36043 Fulda, Germany
Locations (1):
- Kardiologie Lukaskrankenhaus Neuss, Neuss, Germany

REFERENCES:
- [Background] Haude M, Lee SW, Worthley SG, Silber S, Verheye S, Erbs S, Rosli MA, Botelho R, Meredith I, Sim KH, Stella PR, Tan HC, Whitbourn R, Thambar S, Abizaid A, Koh TH, Den Heijer P, Parise H, Cristea E, Maehara A, Mehran R. The REMEDEE trial: a randomized comparison of a combination sirolimus-eluting endothelial progenitor cell capture stent with a paclitaxel-eluting stent. JACC Cardiovasc Interv. 2013 Apr;6(4):334-43. doi: 10.1016/j.jcin.2012.10.018. Epub 2013 Mar 20. PMID 23523459